CLINICAL TRIAL: NCT03997513
Title: The Impact of a Home-based Pulmonary Telerehabilitation Program on Muscle Function and Quality of Life Following Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: The Impact of a Home-based Pulmonary Telerehabilitation Program in Acute Exacerbations of COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F3014-P
Record Dates: First submitted 2019-06-18; First posted 2019-06-25 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: pulmonary disease, chronic obstructive; pulmonary rehabilitation; muscle atrophy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: The intervention will consist of an eight-week, three sessions per week, home-based pulmonary telerehabilitation program that will incorporate both lower extremity endurance exercise and upper and lower extremity resistance training. Subjects randomized to the study intervention will also participate in a one hour, twice-monthly support group via group video conferencing consisting of an educational topic (i.e. inhaler use, understanding COPD) and group discussion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulmonary Telerehabilitation Intervention Group (Experimental): The intervention will consist of an eight-week, three sessions per week, home-based pulmonary telerehabilitation program that will incorporate both lower extremity endurance exercise and upper and lower extremity resistance training. Subjects randomized to the study intervention will also participate in a one hour, twice-monthly support group via group video conferencing consisting of an educational topic (i.e. inhaler use, understanding COPD) and group discussion.
  Interventions: Behavioral: Pulmonary Telerehabilitation
- Usual Care Group (No Intervention): Participants randomized to the usual care arm will also be enrolled in our institution's telehealth program, will receive an automatic blood pressure monitor, portable pulse oximeter, and scale and will be in regular contact with a telehealth provider. A study team member will meet with participants randomized to the usual care arm to discuss the importance of exercise and will encourage exercise (strength training, light aerobic activity such as walking or cycling) a minimum of 20-40 minutes three times per week at discharge.

INTERVENTIONS:
Behavioral: Pulmonary Telerehabilitation — The intervention will consist of an eight-week, three sessions per week, home-based pulmonary telerehabilitation program that will incorporate both lower extremity endurance exercise and upper and lower extremity resistance training. Subjects randomized to the study intervention will also participate in a one hour, twice-monthly support group via group video conferencing consisting of an educational topic (i.e. inhaler use, understanding COPD) and group discussion.
  Arms: Pulmonary Telerehabilitation Intervention Group

SUMMARY:
COPD impacts a significant proportion of the Veteran population. Acute exacerbations, or flare-ups, of COPD are associated with impaired muscle function and worse quality of life. Pulmonary rehabilitation, a formal exercise program for patients with lung disease that includes both endurance and strength training exercises, has been shown to improve muscle function and quality of life after an acute exacerbation of COPD. However, lack of geographically accessible rehabilitation facilities and/or transportation issues are often barriers to pulmonary rehabilitation attendance in the Veteran population. This study will assess the feasibility and impact of an eight-week, three sessions per week, home-based, pulmonary telerehabilitation program in Veterans with COPD following hospitalization for an acute exacerbation of their lung disease. We will measure adherence and satisfaction with the program and muscle strength, physical activity, quality of life, and exercise tolerance pre and post-intervention in Veterans randomized to the pulmonary telerehabilitation arm versus Veterans randomized to the control arm who do not participate in pulmonary rehabilitation.

DETAILED DESCRIPTION:
Pulmonary telerehabilitation programs have been shown to have a high acceptance and adherence rate and lead to improvement in exercise capacity and quality of life in stable COPD. However, data regarding the feasibility and impact of pulmonary telerehabilitation following hospitalization for an Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD) on physical activity levels, muscle function, exercise capacity, and health-related quality of life are lacking. The primary hypothesis is that a home-based pulmonary telerehabilitation program initiated at hospital discharge following an AECOPD is feasible in the Veteran population and will result in increased physical activity and greater improvement in muscle function, exercise capacity, and health-related quality of life compared to usual care. This hypothesis will be tested with the following specific aims: (1) To determine the feasibility of an eight-week home-based pulmonary telerehabilitation program in Veterans with moderate to severe COPD initiated in the immediate post-hospitalization period following an AECOPD. (2) To determine physical activity levels and the magnitude and variability in changes of measurements of muscle strength, functional exercise performance, and health-related quality of life following an eight-week home-based pulmonary telerehabilitation program versus usual care initiated in Veterans with moderate to severe COPD immediately following hospitalization for an AECOPD. The study will randomize (1:1 allocation) 30 male and female Veterans hospitalized with an AECOPD to either an eight-week, three sessions per week, home-based pulmonary telerehabilitation program that includes lower extremity endurance exercises with a cycle ergometer and upper and lower extremity strength training with 1:1 supervision via video conferencing with an exercise physiologist as well as a twice-monthly online support group via video conferencing versus usual care. Changes from baseline in physical activity levels, handgrip and quadriceps muscle strength, exercise endurance, and health-related quality of life will be assessed following the pulmonary telerehabilitation program versus usual care. Findings from this project will contribute to the growing field of pulmonary telerehabilitation and will provide critical preliminary data for the design and implementation of a larger, randomized control trial assessing the impact of pulmonary telerehabilitation on long-term clinical outcomes following AECOPD.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* Moderate or severe COPD with a forced expiratory volume in 1 second - forced vital capacity ratio (FEV1/FVC) < 0.70 and FEV1 < 80% predicted
* Hospitalization with a primary diagnosis of AECOPD, defined as an increase in shortness of breath, cough, and/or sputum production beyond the normal day-to-day variation necessitating a change in regular medication when other causes of increased shortness of breath, cough, and/or sputum production have been ruled out
* Capable of operating a tablet independently with adequate vision and hearing

Exclusion Criteria:

* Acute hypercapneic respiratory failure with a requirement for either non-invasive (i.e. bilevel positive airway pressure) or invasive mechanical ventilation during hospitalization
* Hospitalization < 72 hours
* A secondary diagnosis of acute congestive heart failure, myocardial infarction, or pneumonia during hospitalization or unstable cardiac or neurologic disease at discharge
* Enrollment in a pulmonary rehabilitation program within 12 months of hospitalization
* A medical condition that makes exercise unsafe (includes upper and lower limb strength training and lower limb cycle ergometry)

  * This will be determined by the following- screen for these through chart review, discussion with the patient (do they have any known cardiac issues, do they have chest pain with exertion, are they lightheaded with exertion), discussion with the physicians caring for the patient in the hospital, and direct observation and assessment during the bedside pulmonary rehab sessions (that were built into this study for safety purposes)
* Inclusion in another greater than minimal risk study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Bon Field, MD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pulmonary Telerehabilitation Intervention Group | Usual Care Group
Started | 2 | 3
Completed | 2 | 2
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulmonary Telerehabilitation Intervention Group | Usual Care Group | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2 | 3 | 5
Age, Continuous [Median (Full Range); unit: years] | 68 [65 to 71] | 71 [70 to 75] | 71 [65 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Muscle Strength Testing Change
Description: Quadriceps muscle maximal force (kilogram-force, kgf) will be measured with a Keiser leg press. One repetition maximum (1RM) measures will be obtained by progressively increasing resistance until the participant is unable to successfully complete one repetition. Peak muscle power will be measured at 40, 50, 60, 70, 80, and 90 percent of the 1RM 30 minutes after the 1RM measurement was obtained.
Time Frame: measured at baseline and at ten weeks
Population: This test was not performed due to COVID restrictions at the VA and inability to use the testing equipment.
Arm/Group | Pulmonary Telerehabilitation Intervention Group | Usual Care Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Six Minute Walk Test
Description: Participants completed a six minute walk test, which consisted of walking in a flat corridor for six minutes with the distance walked measured in feet. Participants were instructed to complete the walk using their home oxygen prescription for exertion. The difference between baseline and ten week walk test was compared between groups.
Time Frame: measured at baseline and at ten weeks
Population: One participant in the intervention group declined six minute walk testing at the baseline and follow-up visit. The difference in walk distance from baseline to 10 weeks was compared between groups.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Pulmonary Telerehabilitation Intervention Group | Usual Care Group
Number analyzed (Participants) | 1 | 2
feet | 472 | 48.25 (549.07)

3. Primary Outcome: Health-related Quality of Life Assessments Change
Description: Health-related quality of life will be assessed with the Short-Form 36-Item Questionnaire (SF-36) prior to hospital discharge and at ten weeks following an eight week pulmonary telerehabilitation intervention or usual care. The SF-36 consists of 36 questions spanning nine health domains and is a valid measure of health-related quality of life in COPD that is responsive to change following a pulmonary rehabilitation intervention.
Time Frame: measured at baseline and ten weeks
Population: This questionnaire was not used.
Arm/Group | Pulmonary Telerehabilitation Intervention Group | Usual Care Group
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Participant Satisfaction Survey
Description: Participants will be administered a survey by the study coordinator at ten weeks after completion of the eight-week pulmonary telerehabilitation intervention that will require them to respond to statements related to their satisfaction with the home-based program. Statements will address ease of use of the video conferencing modality, acceptability of exercise components, perceptions of impact on muscle strength and exercise endurance, and willingness to participate in additional pulmonary telerehabilitation. Participants randomized to the usual care group will not be administered a survey.
Time Frame: measured at ten weeks (study completion)
Population: Participants randomized to the pulmonary telerehabilitation intervention group
Measure: Count of Participants; unit: Participants
Arm/Group | Pulmonary Telerehabilitation Intervention Group | Usual Care Group
Number analyzed (Participants) | 2 | 0
Participants
  Participants reporting that exercise sessions were acceptable | 2 |
  Participants reporting tablet interface was easy to navigate once they received instruction on use | 2 |
  Participants reporting adverse events | 0 |
  Participants reporting tolerating exercise well | 2 |

5. Secondary Outcome: Sit-to-stand Test Change
Description: The one-minute sit-to-stand test has been shown to be reliable, valid, and responsive to change in exercise capacity following pulmonary rehabilitation in individuals with COPD. The test consists of the participant standing at full leg extension from a sitting position at their own pace as often as possible during a one minute testing interval. The participant is permitted to stop at any time during the one minute interval if necessary. An armless chair is used for testing and the participant is asked to fold their arms across their chest during testing. Two tests will be performed on separate days prior to discharge and the test with the greatest number of repetitions will be used as the baseline performance measure. A third test will be performed at ten weeks following an eight week pulmonary telerehabilitation intervention or usual care.
Time Frame: measured at baseline and ten weeks
Population: the change in sit to stand count in 30 seconds from baseline to ten weeks between the intervention and usual care group were compared
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | Pulmonary Telerehabilitation Intervention Group | Usual Care Group
Number analyzed (Participants) | 2 | 2
repetitions | 9.5 (6.4) | 5 (1.4)

6. Secondary Outcome: Handgrip Strength
Description: Handgrip strength of the dominant hand will be measured with a hand dynamometer. Three measurements will be taken with a 60 second recovery period between trials. The average maximal force across trials will be calculated as the final handgrip strength.
Time Frame: measured at baseline and ten weeks
Population: change in handgrip strength from baseline to ten weeks compared between groups
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Pulmonary Telerehabilitation Intervention Group | Usual Care Group
Number analyzed (Participants) | 2 | 2
Kg | 1.75 (3.18) | 0.5 (12.02)

7. Secondary Outcome: Disease Specific Quality of Life
Description: The St. George's Respiratory Questionnaire (SGRQ) is a disease-specific questionnaire validated to measure health status in patients with COPD. Total SGRQ scores range from 0-100 with higher scores indicating greater symptoms burden. The minimal clinically important difference is a difference of four points in the total SGRQ score.
Time Frame: measured at baseline and ten weeks
Population: change in SGRQ score from baseline to ten weeks compared between groups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulmonary Telerehabilitation Intervention Group | Usual Care Group
Number analyzed (Participants) | 2 | 2
score on a scale | -.19 (20.9) | -17.8 (4.3)

8. Secondary Outcome: Symptoms During Sit-to-stand Test
Description: The participants' perception of dyspnea and exertion during the sit-to-stand test will be assessed following each test with the ten point Borg dyspnea and leg fatigue scale, which measures the degree of dyspnea and leg fatigue with exercise.
Time Frame: measured at baseline and ten weeks
Population: not systematically assessed during the study
Arm/Group | Pulmonary Telerehabilitation Intervention Group | Usual Care Group
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Post-intervention Survey
Description: Questions regarding social support, psychiatric attributes, and other factors potentially associated with program adherence will be asked in order to gain preliminary insights to optimize recruitment for a larger, randomized controlled trial of pulmonary telerehabilitation.
Time Frame: measured at ten weeks (study completion)
Population: Not administered.
Arm/Group | Pulmonary Telerehabilitation Intervention Group | Usual Care Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from signed consent until completion of either the intervention or usual care group, which was a period of 12-14 weeks.
Arm/Group | Pulmonary Telerehabilitation Intervention Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

LIMITATIONS AND CAVEATS:
The study was significantly impacted by the COVID-19 pandemic due to months of restrictions on human subject research and national trends of fewer hospitalized acute exacerbations of COPD as seen in the COPD population during the height of the pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT03997513/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT03997513/ICF_000.pdf